CLINICAL TRIAL: NCT02352194
Title: Observational Study of the Physical Capacity of Patients With Multiple Sclerosis and Evaluation of the Effects of Usual Rehabilitation in the Day Hospital
Brief Title: Physical Capacity and Rehabilitation of Patients With Multiple Sclerosis
Acronym: REHABSEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 14-REHABSEP
Record Dates: First submitted 2015-01-20; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple Sclerosis, Physical therapy, Physical capacity, Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Assessment: One part of this study is to quantify physical capacity of patients with Multiple sclerosis.
  Thirty patients will be enrolled in this study and performed assessments.
- Rehabilitation: A second part of this study is to quantify the benefit of a usual rehabilitation program in the day hospital. Thirty patients will be enrolled in this study and receive rehabilitation. They will be assessed before and after the rehabilitation program (physiotherapy and physical activity)
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Physiotherapy and physical activity
  Groups: Rehabilitation

SUMMARY:
The purpose of this study is to assess the physical capacity of patients with multiple sclerosis and the effects of rehabilitation, encompassing physical therapy and physical activity as it is carried out in the day hospital of (the Physical and Rehabilitation Medicine department) at Garches Hospital. We will compare the results of assessments carried out before and after a standard rehabilitation program.

DETAILED DESCRIPTION:
Single center, retrospective and prospective study.

In order to assess the efficiency of the of usual rehabilitation proposed to patients in the day hospital, assessments are systematically performed before and after the rehabilitation program:

1. Assessment of muscular strength and fatigue:

   Assessments of voluntary force will be those usually performed in the context of the evaluation of patients. The isokinetic dynamometer CON-TREX ® is a device that provides a quantified result of the torque developed in a predetermined joint area with a constant speed which is also defined in advance.

   The assessment includes an assessment of the strength in isometric contraction (at 40 and 90 degrees of knee flexion) and concentric contraction (30, 60 and 90 degrees per second). Fatigue is evaluated by two self-administered questionnaires: the Fatigue Severity Scale and Modified Fatigue Impact Scale.
2. Effort test:

   The aerobic capacity of patients will be assessed by a triangular maximal exercise test.

   The effort test is performed on a cycle ergometer from a triangular incremental exercise. Beforehand, blood pressure and ECG are recorded to establish that the patient can safely achieve a gradual stress test. Heart rate, blood pressure, oxygen consumption, the feeling (Borg scale) and ECG are recorded immediately before and immediately after the end of the test and every minute for at least 5-10 minutes during the recovery phase.
3. Clinical assessment:

The Timed Up and Go test will be used to assess the patient's capacity of postural transition.

This is a timed quantitative assessment of the duration needed to change from sitting in a chair, get up and walk three meters, make a U-turn and come back to sit down.

The 10 meters test quantifies the walking speed of patients (meters / second) over 10 meters A test of ascending and descending10 stairs is also performed, as well as the 6 minutes walking test.

In addition to these functional assessments, clinical tests are conventionally performed such as the measurement of muscle strength (Medical Research Council scale), range of motion, spasticity (modified Ashworth scale) and an assessment of the balance and posture.

The SEP-59 questionnaire will be used to assess the patients quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis with EDSS ≤ 6 (Expanded Disability Status Scale)
* Patient ≥ 18 years old
* Patient able to comply with the recommended monitoring
* No relapse within the last three months
* More than six months elapsed since last medical care in day hospital
* No recent modification (six month) of medications for MS
* More than three months elapsed since last change of associated treatments (Fampyra, botulinum toxin)

Exclusion Criteria:

* Patients under any form of guardianship or curatorship
* Breastfeeding
* Orthopedic complications with repercussions on walking activities
* No affiliation to a social security scheme (beneficiary or assignee)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with MS since at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the strength and fatigue | Within 10 weeks from the start of the rehabilitation program
  Assessment realised with an isokinetic dynamometer

SECONDARY OUTCOMES:
6 minutes walking test | Within 10 weeks from the start of the rehabilitation program
  Patients were instructed to walk as far as possible in a 50 meters corridor during 6 minutes
Evaluation of aerobic capacity during an effort test | Within 10 weeks from the start of the rehabilitation program
  Aerobic capacity (VO2max)
Assessment of the balance of patients | Within 10 weeks from the start of the rehabilitation program
  Berg Balance Scale
Assessment of Spasticity with the Modified Ashworth Scale (MAS), | Within 10 weeks from the start of the rehabilitation program
10 meters Walk test | Within 10 weeks from the start of the rehabilitation
  Patients have to walk over a 14 meter walkway and time required to traverse the middle 10 meters of the walk was recorded to avoid acceleration and deceleration effects
Timed up and go test | Within 10 weeks from the start of the rehabilitation
  Patients have to get up from a chair, walk 3 meters, turn around and return to sitting as quickly as possible
Time to ascend and descend stairs | Within 10 weeks from the start of the rehabilitation
  Participants were instructed to ascend and descend 10 stairs using the hand rail
Assessment of Strength with the Medical Research Council (MRC), | Within 10 weeks from the start of the rehabilitation
Assessment of Quality of Life with SEP-59 Scale | Within 10 weeks from the start of the rehabilitation
Assessment of the balance of patients | Within 10 weeks from the start of the rehabilitation
  Postural control assessment : eyes opened and eyes closed

CONTACTS AND LOCATIONS:
Overall Officials: Djamel Bensmail, MD,PhD, Principal Investigator — Physical and Rehabilitation Medicine department, Raymond Poincaré Hospital,; Raphael Zory, PhD, Study Director — LAMHESS Laboratory, Faculty of Sports Science, 06205 Nice, France; Sophie Hameau, Study Director — Physical and Rehabilitation Medicine department, Raymond Poincaré Hospital,
Locations (1):
- Raymond Poincaré Hospital, Garches, France

REFERENCES:
- [Derived] Hameau S, Bensmail D, Roche N, Zory R. Fatigability in Patients With Multiple Sclerosis During Maximal Concentric Contractions. Arch Phys Med Rehabil. 2017 Jul;98(7):1339-1347. doi: 10.1016/j.apmr.2016.12.014. Epub 2017 Jan 25. PMID 28130080